CLINICAL TRIAL: NCT05615129
Title: Effect of Immunochemotherapy Sequence and Time-of-day Infusion on Efficacy and Prognosis of Patients With Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Sequence and Time-of-day Infusion of immunoCHemotherapy Affect Response in Oesophageal Cancer in the NeOadjuvant Setting
Acronym: RICE-Chronos
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital of Shantou University Medical College (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RICE-Chronos
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is reported that compared to chemotherapy alone, immunochemotherapy has significantly improved the overall survival of patients with advanced metastatic ESCC. However, there are still more than 30% of patients who cannot benefit from this treatment modality. In addition to these factors, the time-of-day infusion and administration sequence of immunochemotherapy have been reported to be associated with tumor responses and overall survival. In this study, The investigators aimed to explore the roles of infusion time and administration sequence of immunochemotherapy in predicting tumor responses and overall survival in patients with advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as esophageal squamous cell carcinoma
* KPS≥80
* Adequate organ function
* No distant metastasis
* The diseases could be resected or potentially resectable after immunochemotherapy assessed by a thoracic oncologist

Exclusion Criteria:

* incomplete medical record which affects statistical analysis
* have participated in previous interventional clinical trials
* other situations evaluated by investigators not meet the enrollment

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as potentially resectable (including initially-unresectable) esophageal squamous cell carcinoma via pathological specimen, KPS ≥ 80, has adequate organ function and no distant metastasis are included in the study
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | from the date of diagnosis to the date of death, assessed up to 100 months
  Overall survival rate

SECONDARY OUTCOMES:
Pathologic complete response rate (pCR) | Three to five working days after surgery
  The rate of pathologic complete response rate after the combined treatment of chemotherapy and immunotherapy following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China